CLINICAL TRIAL: NCT01513330
Title: An Open-labelled, Randomised, Controlled, Crossover Investigation Evaluating Performance of a Newly Developed Ostomy Care Product Compared to Standard Care.
Brief Title: Performance Study of Newly Developed Ostomy Products
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Coloplast A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: CP219
Record Dates: First submitted 2012-01-10; First posted 2012-01-20 (Estimated); Results first posted 2014-01-09 (Estimated); Last update posted 2014-01-09 (Estimated); Status verified 2013-11

CONDITIONS: Stoma Colostomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- First Standard Care, then SenSura Mio (Experimental): Subjects first test Standard Care (Either SenSura, Nova 1, Moderna/Moderna Flex, Esteem or Flexima/Softima) and after cross-over SenSura Mio
  Interventions: Device: SenSura Mio; Device: Standard Care
- First SenSura Mio, then Standard Care (Experimental): Subjects first test SenSura Mio and after cross-over Standard Care(Either SenSura, Nova 1, Moderna/Moderna Flex, Esteem or Flexima/Softima)
  Interventions: Device: SenSura Mio; Device: Standard Care

INTERVENTIONS:
Device: SenSura Mio — Ostomy product - 1 piece closed bag
Device: Standard Care — Ostomy product 1 piece closed bags. Either SenSura, Nova 1, Moderna/Moderna Flex, Esteem or Flexima/Softima.

SUMMARY:
The purpose of the study is to evaluate leakage of a newly developed ostomy product compared to standard care in subjects with colostomies. Subjects will be asked to use each test product for 2 weeks - in total, the study period is 4 weeks and the hypothesis is to show that the newly developed ostomy product is significantly better to reduce leakage compared to standard care.

ELIGIBILITY:
Inclusion Criteria:

1. Have given written informed consent.
2. Be at least 18 years of age and have full legal capacity.
3. Have experienced leakage under the base plate at least once a week over the last two weeks.
4. Be able to handle the bags themselves or with help from caregiver (e.g. spouse).
5. Have a colostomy with a diameter between 20 and 45 mm.
6. Have had their ostomy for at least three months.
7. Currently use a 1-piece flat product with closed bag.
8. Use minimum 1 product per day.
9. Be suitable for participation in the investigation and for using a standard adhesive, flat base plate (evaluated by investigator).

Exclusion Criteria:

1. Use irrigation during the study (flush the stoma with water).
2. Currently receiving or have within the past 2 months received radio- and/or chemotherapy.
3. Currently receiving or have within the past month received local or systemic steroid treatment in the peristomal area.
4. Are pregnant or breastfeeding.
5. Participating in other interventional clinical investigations or have previously participated in this investigation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2011-11; Primary Completion 2012-06 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wenche Sundberg, stoma nurse, Principal Investigator — Diakonhjemmet Sykhus, Oslo; Merete Bjørke, Stoma Nurse, Principal Investigator — St. Olavs Hopsital; Vigids Dagsland, Stoma Nurse, Principal Investigator — Haugesund Sykhus; Randi Melum, Stoma Nurse, Principal Investigator — St. Olavs Hospital
Locations (1):
- Publicare, Cologne, Køln, Germany

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The subjects were recruited via sites and user data-bases in Denmark, Norway, Germany and France.
Groups:
- First SenSura Mio, Then Standard Care: The subjects first test SenSura Mio : Ostomy product - 1 piece closed bag and thereafter cross-over and test Standard Care (Either SenSura, Nova 1, Moderna/Moderna Flex, Esteem or Flexima/Softima)
- First Standard Care, Then SenSura Mio: The subjects first test Standard Care Ostomy product 1 piece closed bags (Either SenSura, Nova 1, Moderna/Moderna Flex, Esteem or Flexima/Softima)and after cross-over test SenSura Mio 1-piece closed bags.
Period: SenSura Mio First,
Arm/Group | First SenSura Mio, Then Standard Care | First Standard Care, Then SenSura Mio
Started | 64 | 58
Completed | 60 | 56
Not Completed | 4 | 2
Not completed — Adverse Event | 2 | 0
Not completed — Lack of Efficacy | 0 | 1
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Other | 1 | 0
Period: Standard Care First,
Arm/Group | First SenSura Mio, Then Standard Care | First Standard Care, Then SenSura Mio
Started | 60 | 56
Completed | 56 | 52
Not Completed | 4 | 4
Not completed — Lack of Efficacy | 2 | 2
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Other | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: Entire study population = all participants enrolled in the study
Arm/Group | Entire Study Population
Number analyzed (Participants) | 122
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.3 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 63
  Male | 59

OUTCOME MEASURES:

1. Primary Outcome: Degree of Leakage. Each Baseplate Can Have a Score From 0-24 Points Were 0 is the Best Possible Outcome (No Leakage) and 24 Points is the Worst Possible Outcome (Full Plate Leakage)
Description: Degree of leakage will be measured by a 25-point leakage scale (no leakage or up till 24 points of leakage), developed by Coloplast A/S. The subjects receive Petri dishes with pre-printed leakage scale on. The subject will place the Petri dish above the used baseplate and indicate where on the baseplate output appears. This is done by ticking of each area on the scale indicating the area of leakage.
Time Frame: 14 days
Measure: Mean (Standard Deviation); unit: points on a scale
Units Other Than Participants: baseplates
Groups:
- SenSura Mio: SenSura Mio : Ostomy product - 1 piece closed bag
- Standard Care: Standard Care : Ostomy product 1 piece closed bags. Either SenSura, Nova 1, Moderna/Moderna Flex, Esteem or Flexima/Softima.
Arm/Group | SenSura Mio | Standard Care
Number analyzed (Participants) | 120 | 118
Number analyzed (baseplates) | 2852 | 2810
points on a scale | 3.8 (5.0) | 3.4 (4.4)

ADVERSE EVENTS:
Arm/Group | SenSura Mio | Standard Care
Serious Adverse Events (participants affected / at risk) | 0/120 | 0/118
Other Adverse Events (participants affected / at risk) | 10/120 | 10/118
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SenSura Mio (N=120) | Standard Care (N=118)
Itching (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Peristomal skin redness (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3)
Peristomal skin erosion (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Peristomal allergic contact dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) — Not clinically verified allergic contact dermatitis.1 subject tested 21 Nova baseplates before the AE -allergic dermatitis.1 subject tested 8 SenSura Mio baseplates during 3 days before the AE -contact dermatitis because of allergic reaction occured.
Peristomal burns (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (2) | 0 (0)
Infected toe (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Consumption of food leading to skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Granulation in the peristomal area (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Pain in the peristomal area (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No